CLINICAL TRIAL: NCT06211504
Title: Sinus Tarsi Implant as an Adjuvant Procedure to Medial Displacement Calcaneal Osteotomy in the Treatment of Mobile Adult Acquired Flatfoot Deformity: a Randomized Controlled Trial
Brief Title: Sinus Tarsi Implant as an Adjuvant Procedure to Medial Displacement Calcaneal Osteotomy in the Treatment of Mobile Adult Acquired Flatfoot Deformity
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-02892-01
Record Dates: First submitted 2023-11-13; First posted 2024-01-18 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Acquired Adult Flatfoot Deformity; Flat Foot; Flexible Flatfoot
Keywords: AAFD; RCT; clinical trial; surgical intervention; arthroereisis; sinus tarsi implant
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- MDCO without STI (Active Comparator): 1. For patients with preoperative gastrocnemius-soleus complex tightness, defined as a preoperative dorsal extension of the ankle less than 5 degrees, with the knee completely extended, a Strayer´s procedure will be performed before the other procedures.
  2. MDCO will be performed where the distal aspect of the calcaneus is separated from the proximal aspects, slided medially and fixed with two screws.
  3. After the MDCO, FDL will be transferred to the navicular bone.
  4. The spring ligament will be assessed. If ruptured, it will be reconstructed. If not ruptured, it will be tightened.
  5. A plantarflexing open wedge osteotomy of the medial cuneiform (Cotton osteotomy) will be performed if pre-/perioperative findings indicate it.
  Interventions: Procedure: Conventional surgery
- MDCO with STI (Experimental): 1. In patients with preoperative gastrocnemius-soleus complex tightness, defined as a preoperative dorsal extension of the ankle less than 5 degrees, with the knee completely extended, a Strayer´s procedure will be performed before the other procedures.
  2. Thereafter, an STI (ProStop® Arthroereisis Subtalar Implant, Arthrex GmbH, Munich, Germany) will be inserted into the sinus tarsi.
  3. MDCO will be performed where the distal aspect of the calcaneus is separated from the proximal aspects, slided medially and fixed with two screws.
  4. After the MDCO, FDL will be transferred to the navicular bone.
  5. The spring ligament will be assessed. If ruptured, it will be reconstructed. If not ruptured, it will be tightened.
  6. A plantarflexing open wedge osteotomy of the medial cuneiform (Cotton osteotomy) will be performed if pre-/perioperative findings indicate it.
  Interventions: Device: ProStop, sinus tarsi implant (STI); Procedure: Conventional surgery

INTERVENTIONS:
Device: ProStop, sinus tarsi implant (STI) — Insertion of a sinus tarsi implant (ProStop from Arthrex) in sinus tarsi
  Other Names: arthroereisis
  Arms: MDCO with STI
Procedure: Conventional surgery — MDCO - medial displacement calcaneal osteotomy FDL transfer - flexor digitorum longus tendon transfer to the navicular bone Spring ligament repair - reconstruction of the spring ligament Strayer's procedure - gastrocnemius recession (if necessary) Cotton osteotomy - medial cuneiform opening wedge osteotomy (if necessary)

SUMMARY:
Background: Adult acquired flatfoot deformity (AAFD) is a deformity of the foot which leads to pain and an altered gait pattern. There are several different surgical interventions available for treatment of AAFD. One of the most common treatments for mobile AAFD is medial displacement calcaneal osteotomy (MDCO) with or without adjuvant soft tissue procedures. However, the medial displacement of the calcaneus only aims to correct the deformity in one plane despite AAFD being a deformity of three planes with hypereversion of the calcaneus, anterior translation of the talus over the calcaneus and tilting/drop of the calcaneal head. Because of these multiple forces, the healing of MDCO in the intended position can sometimes be hard to achieve and medial soft tissue is still stressed leading to recurring deformity. The investigators believe that adjuvant insertion of a sinus tarsi implant (STI) could work as an internal splint, protecting soft tissue procedures on the medial side, reversing anterior translation of the talus, opposing calcaneus eversion, and lifting talar head. This additional procedure will create a better correction of the deformity with enhanced appearance of the foot and better long-term functional results.

Methods: This is a multi-center randomized controlled trial designed to assess the efficacy of STI as an adjuvant procedure to MDCO in patients with mobile AAFD (Stage II). Patients aged 16 to 75 years, referred to one of the orthopedic centers involved in this study, will be invited to participate if they fulfil the trials eligibility criteria. In total, 130 patients who provide informed consent will be randomized to either MDCO with STI or MDCO without STI (65 patients in each group). The included patients will be clinically and radiographically examined. They will also fill out a form before surgery and 4-5 months, 1 year and 2 years postoperatively. The form will include Self-Reported Foot and Ankle Score (SEFAS) and Euro-QoL 5 Dimensions (EQ-5D). The trials primary outcome will be change in Meary's angle. Secondary outcomes include additional radiographic changes, change in SEFAS score, EQ-5D index, pain according to visual analog scale (VAS), satisfaction assessment, clinical outcome measures, the length of postoperative sick-leave and rate of complications.

Discussion: This is the first randomized controlled trial assessing the efficacy of a sinus tarsi implant as an adjuvant procedure to MDCO.

DETAILED DESCRIPTION:
MDCO is a commonly used procedure with few complications. However, the medial displacement of the calcaneus only aims to correct the deformity in one plane despite AAFD being a deformity of three planes with hypereversion of the calcaneus, anterior translation of the talus over the calcaneus and tilting/drop of the calcaneal head. Because of these multiple forces, the healing of MDCO in the intended position can sometimes be difficult to achieve and medial soft tissue is still stressed leading to recurring deformity. The sinus tarsi implant (STI) has been described to function as an internal splint, protecting soft tissue procedures on the medial side, reversing anterior translation of the talus, opposing calcaneal eversion, and lifting talar head. This is suggested to create a better correction of the deformity with enhanced appearance of the foot and potentially better long-term functional results.

Methods

Trial design and setting The study is a prospective multicenter randomized controlled trial conducted at nine orthopedic centers in Sweden. The participating centers are Hässleholm hospital, Skåne University Hospital in Malmö, Capio Ortho Center in Malmö and Göteborg, Sahlgrenska University hospital in Mölndal, Uppsala University Hospital, Falun Hospital, Östersund Hospital, Eksjö Hospital and Växsjö Hospital.

Screening

Patients referred to the orthopedic department at the participating centers will be evaluated by an orthopedic specialist with history and clinical examination. There will usually be radiographic imaging done before the visit. With clinical and radiographic examination, the surgeon can usually establish a diagnosis of AAFD and decide whether surgical treatment is indicated. Patients judged to fulfil the eligibility criteria are then given, by the surgeon, full verbal and written information about the aims and conduct of the trial as well as potential advantages and disadvantages of participation. Patients who accept participation will provide written informed consent.

Patients who consent to participate will undergo baseline assessment at another appointment scheduled between the screening and the date of surgery.

Randomization

Patients are centrally randomized according to a computer-generated randomization list (ratio 1:1). The randomization is stratified according to patient sex and is done in random blocks of various sizes.

Follow-up procedures

Patients will complete a questionnaire consisting of two PROMs, the generic EuroQol 5 Dimensions (EQ-5D) and the Self-reported Foot and Ankle Score (SEFAS) as well as 5 additional questions regarding how pleased (satisfied) the patients are with the appearance of the foot, the shoes they are able to wear, foot strength, stability, and their overall satisfaction with the results of the surgery (this question will be included in the postoperative questionnaire). The questionnaires will be completed at baseline, 4-5, 12, and 24 months postoperatively. At these follow-up visits, the patients will also be clinically examined by a physiotherapist or nurse, and radiographic examination will be done. The trial coordinator will monitor completeness of questionnaires and use telephone contact when necessary. Participants are informed, in writing and during examination/follow-up, about the importance of completing the follow-up questionnaires and examinations. Patients can choose to discontinue study participation at any given time point without being obliged to an explanation.

Outcome measures

Changes in the alignment of the foot will be assessed with weight-bearing radiographs measuring specific angles and positions described below.

The EQ-5D is a validated generic PROM that assess health status and health-related quality of life from 5 different dimensions. The 5 dimensions are summarized in an index where 1 represents best health status and 0 the lowest health status. In the EQ-5D, the patient can also estimate their general health on a scale from 0 to 100 on a visual analog scale (VAS). EQ-5D sex-specific, country-specific, and age-specific normative values are available, which makes comparison between a healthy population and the study participants possible.

Self-reported Foot and Ankle Score (SEFAS) is a foot- and ankle-specific PROM based on the New Zealand total ankle questionnaire (NZAQ) and the Swedish version has been created according to a standardized cross-cultural adaption procedure. The PROM contains different dimensions including pain, function, and activity limitations. The different dimensions are summarized into a total score where 0 represents most severe disability and 48 represents normal function. A system has been created for handling of incorrect completion or missing answers in the SEFAS. The SEFAS has been validated for foot and ankle disorders. Gender- and age-specific normative values have also been collected for the Swedish population and the minimal important change (MIC) value have been calculated for SEFAS. A change in SEFAS score of 5 units is considered clinically relevant.

Pain will be measured with a visual analog scale (VAS) asking the patients to rate (on 0 to 100 scale) their pain severity.

Satisfaction will be assessed with five additional questions on a five item Likert scale:

1. How satisfied is the participant with the appearance of his/her foot?
2. How satisfied is the participant with the shoes he/she is able to wear?
3. How satisfied is the participant with the strength of the foot?
4. How satisfied is the participant with the stability of the foot?
5. How satisfied is the participant with the results of the surgery (not applicable at baseline assessment)? The participants will also answer a question about the duration of postoperative sick leave in the postoperative questionnaires.

Physical examination

The physical examinations will be performed by a physiotherapist or a nurse and will include evaluation of single heel-rise height (cm from the lowest part of the heel to the floor) and endurance (number of performed heel-rises). The examiner will be blinded to group allocation and steristrips will be placed in front of the lateral malleolus in order to cover surgical scars that may be located there.

Radiographic examination Meary's angle is the angle between the midline of talus and the midline of the first metatarsal bone on a lateral view radiograph. In a normally configurated foot this angle is approximately 0 degrees. In the flatfoot, talus frontal portion collapses towards the floor which increases Meary's angle that becomes greater the more talus collapses downward. Radiographic examination will include foot and ankle (frontal projection and from the side) at weight-bearing.

Presence of malalignment of the ankle fork will be noted from the frontal projection of the ankle and the Salzman view. CT or MRI will not be performed pre- or postoperatively if there is no specific reason, in that case, reported by the treating surgeon.

Adherence

In written information, before randomization, and during all contacts with the research team the trial participants will be informed about the importance of remaining in the trial, completing the questionnaires, and participating in the follow-up examinations.

Postoperative regimes Patients will receive external fixation in the form of a cast postoperatively. Patients who have undergone Cotton osteotomy will wear the cast for 8 weeks postoperatively and will not be allowed to bear weight on the operated foot for three weeks postoperatively. Patients who have not undergone a Cotton osteotomy will wear the cast for 6 weeks postoperatively and will bear weight on the operated side immediately postoperatively. When the patients start bearing weight postoperatively, they will use crutches for support.

Surgery

Surgery will be done by experienced foot and ankle surgeons, defined as orthopedic specialists (senior consultants) with at least 15 forefoot and/or 5 hindfoot procedures yearly, at the participating centers.

Assessment of safety

During the conduct of the trial, the investigator will report all adverse events. All adverse events will be followed up until resolved or as clinically required. Adverse events may be reported spontaneously by the patient or elicited through open questioning during and at the end of the trial. Participants are informed to contact the trial therapists or coordinator at the participating centers whenever they wish to discuss or report any events during the trial period. All reported or observed adverse events including type, intensity and duration will be recorded in a standard protocol. Any serious adverse events will be promptly reported to the steering and data monitoring committees and the trial sponsor. Extraction of the STI due to pain/discomfort or other reason will be monitored and reported but not considered an adverse event or a reason for termination of the trial.

Assessment of costs

The investigators will assess the cost-effectiveness of the respective procedures by comparing duration of surgery, material costs, complication rate and potential need of additional health-care visits or procedures.

Withdrawals Patients can withdraw from the trial at any time without need to give reasons. Patients who do not wish to attend physical examination will be asked to complete the questionnaire.

Sample size

The primary outcome is change in Meary's angle from baseline to 1 year postoperatively. In previous studies investigating the degree of correction in Meary's angle from baseline to 1 year after MDCO in patients with AAFD stage IIa, a mean correction of 10 degrees has been reported.

Assuming a mean correction of Meary's angle of 10 degrees (SD 10) after MDCO and 15 degrees (SD 10) after MDCO with an adjuvant STI, 80% power and p<0.05, a sample size of 63 patients in each trial arm will be required. The investigators aim to recruit 130 patients (65 in each treatment group) because of potential dropouts.

Statistical analysis

For continuous endpoints (radiographic measurements, SEFAS score, EQ-5D index, heel-rise height and endurance, duration of sick-leave) mean values and standard deviations will be calculated. For categorical variables, such as adverse events, and satisfaction assessment, proportions will be calculated. Statistical tests will be performed according to the intention-to-treat principle. An exploratory as-treated analysis will also be performed.

Both hypothesis-generating and confirmatory testing will be performed, the latter for the primary endpoints.

Primary analysis: The mean degree change in Meary's angle from baseline to 12 months postoperative (primary outcome) will be compared using paired samples t-test.

Secondary analyses:

Mean change in residual radiographic measurements, SEFAS score and EQ5D index, clinical tests, duration of sick-leave will be investigated using paired samples t-test. Adverse events and satisfaction assessment will be presented in tables.

Missing values

For the patient-reported measures missing item responses will be managed according to the instructions specific to each scale. If number of missing items precludes calculating a score, the missing score will not be replaced. Missing values for other variables will not be replaced.

Blinding

Patients will be blinded to what surgical procedure will be performed. The primary outcome is radiographic changes in Meary's angle. Follow-up clinical examinations will be done by blinded assessors by placing steristrips in front of lateral malleolus that will cover scars from the surgical procedures prior to examination. The radiographic measurements will be performed by two external radiologists blinded to group allocation. Prior to radiographic assessment, the radiographs will be masked by a person not involved in the assessment, using a computer program covering the place where an STI could be placed (provided it does not interfere with accurate measurement of Meary's angle).

All statistical analyses will be done by a statistician blinded to group allocation.

Ethics

The trial will be conducted in accordance with the declaration of Helsinki. The project has been examined and received approval by the Swedish Ethical Review Authority (Dnr 2023-02892-01 and DNR 2025-05078-02).

Recruitment strategy and timeline

The 10 included orthopedic centers involved in this trail have an AAFD surgery rate of 4 to 20 per year. The investigators aim to recruit 130 patients (65 in each treatment group) and estimate the recruitment of patients will take approximately 2 years.

Patients will be asked to participate according to the screening process described above.

Discussion

Previous studies have shown low health-related quality of life (HRQoL) prior to surgery in patients with AAFD. A postoperative improvement in HRQoL and measured radiographic deformity have been shown for many surgical interventions including MDCO. However, the radiographic improvement has been shown to diminish progressively after surgery and many patients must be treated surgically again.

The STI has been used for many years as a single intervention or adjuvant procedure in the treatment of AAFD. However, the evidence regarding its effect is limited. There are a few studies suggesting an added radiographic improvement when the STI is used as an adjuvant procedure, but to confirm these findings higher-quality evidence is needed. In this trial, the investigators aim to assess the results of STI as an adjuvant procedure to MDCO in the treatment of AAFD stage IIa compared to conventional treatment. The investigators believe this study can generate high-level evidence in an area where current evidence is lacking. If an additive effect of the STI can be proven, it may lead to change in clinical practice and improve the quality of life and foot function in patients suffering from AAFD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AAFD stage II, in whom the talonavicular uncoverage is not considered by the treating surgeon to require an additional lateral column lengthening
* Age 16-75 years, either sex
* Failed non-surgical treatment including 3 months of physiotherapy

Exclusion Criteria:

* Previous ipsilateral surgery for AAFD
* General hypermobility (Beighton score > 6)
* Osteoarthritis in the hindfoot joints, ankle joint or first tarsometatarsal joint
* Rheumatoid arthritis
* Inability to answer patient-reported outcome measures (PROMs) due to language difficulties or cognitive disorder
* Current smoker
* Current pregnancy
* Severe medical illness
* Known abuse of drugs and/or alcohol
* Previous ipsilateral hindfoot fracture including Lisfranc injury

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Meary's angle | From baseline/preoperatively (max 6 months preoperatively) to 12 months postoperatively
  Change in degrees of Meary's angle

SECONDARY OUTCOMES:
Meary's angle | From baseline/preoperatively (max 6 months preoperatively) to 4-5 and 24 months postoperatively
  Change in degrees of Meary's angle
Calcaneal inclination angle | From baseline/preoperatively (max 6 months preoperatively) to 4-5, 12, and 24 months postoperatively
  Change in degrees of Calcaneal inclination angle
Talar declination angle | From baseline/preoperatively (max 6 months preoperatively) to 4-5, 12, and 24 months postoperatively
  Change in degrees of talar declination angle
Talar-2nd metatarsal angle | From baseline/preoperatively (max 6 months preoperatively) to 4-5, 12, and 24 months postoperatively
  Change in degrees of talar-2nd metatarsal angle
Talar coverage angle | From baseline/preoperatively (max 6 months preoperatively) to 4-5, 12, and 24 months postoperatively
  Change in degrees of talar coverage angle
Talar uncoverage | From baseline/preoperatively (max 6 months preoperatively) to 4-5, 12, and 24 months postoperatively
  Change in percentage of talar uncoverage
Medial cuneiform height | From baseline/preoperatively (max 6 months preoperatively) to 4-5, 12, and 24 months postoperatively
  Change in height of the medial cuneiform bone to the floor
Angle between tibial and calcaneal midline | From baseline/preoperatively (max 6 months preoperatively) to 4-5, 12, and 24 months postoperatively
  Change in degrees of the angle between tibial and calcaneal midline on Salzman view
SEFAS change | From baseline/preoperatively (max 6 months preoperatively) to 4-5, 12, and 24 months postoperatively
  Change in Self-Reported Foot and Ankle Score (0-48), where 0 represents worst function and pain in the foot and 48 represent normal function without pain
EQ5D-3L change | From baseline/preoperatively (max 6 months preoperatively) to 4-5, 12, and 24 months postoperatively
  Change in the 3-level version of EuroQol-5-Dimension index (0-1), where 0 represents worst possible general health status of the patient and 1 represents best possible health status
VAS change | From baseline/preoperatively (max 6 months preoperatively) to 4-5, 12, and 24 months postoperatively
  Change in visual analog scale where 0 represents no pain and 10 represents worst possible pain
Degree of satisfaction regarding the results of the surgery | Measured at 4-5, 12, and 24 months postoperatively
  A question "How satisfied are you with the results of the surgery?" will be answered with one of five options: 1. "Very satisfied", 2. "Satisfied", 3. "Quite satisfied", 4. Neither satisfied nor unsatisfied", 5. "Dissatisfied"
Degree of satisfaction regarding the appearance of foot | From baseline/preoperatively (max 6 months preoperatively) to 4-5, 12, and 24 months postoperatively
  A question "How satisfied are you with the appearance of your foot?" will be answered with one of five options: 1. "Very satisfied", 2. "Satisfied", 3. "Quite satisfied", 4. Neither satisfied nor unsatisfied", 5. "Dissatisfied"
Degree of satisfaction regarding the shoe-wear | From baseline/preoperatively (max 6 months preoperatively) to 4-5, 12, and 24 months postoperatively
  A question "How satisfied are you with the shoes you are able to wear?" will be answered with one of five options: 1. "Very satisfied", 2. "Satisfied", 3. "Quite satisfied", 4. Neither satisfied nor unsatisfied", 5. "Dissatisfied"
Degree of satisfaction regarding the strength of the foot | From baseline/preoperatively (max 6 months preoperatively) to 4-5, 12, and 24 months postoperatively
  A question "How satisfied are you with the strength of your foot?" will be answered with one of five options: 1. "Very satisfied", 2. "Satisfied", 3. "Quite satisfied", 4. Neither satisfied nor unsatisfied", 5. "Dissatisfied"
Degree of satisfaction regarding the stability of the foot | From baseline/preoperatively (max 6 months preoperatively) to 4-5, 12, and 24 months postoperatively
  A question "How satisfied are you with the stability of your foot?" will be answered with one of five options: 1. "Very satisfied", 2. "Satisfied", 3. "Quite satisfied", 4. Neither satisfied nor unsatisfied", 5. "Dissatisfied"
Adverse events | At 12 and 24 months postoperative
  Number of adverse events
Single heel-rise peak height | From baseline/preoperatively (max 6 months preoperatively) to 4-5, 12, and 24 months postoperatively
  Change in single heel-rise peak height (cm from lowest part of heel to floor)
Single heel-rise endurance | From baseline/preoperatively (max 6 months preoperatively) to 4-5, 12, and 24 months postoperatively
  Change in single heel-rise endurance (total positive work)
Length of sick-leave | Asked at 4-5, 12 and 24 months postoperative
  Duration of postoperative sick-leave

CONTACTS AND LOCATIONS:
Overall Officials: Ida Osbeck, MD, Principal Investigator — Region Skane
Locations (10):
- Sweden (10):
  - Department of Orthopedics - Hässleholm Hospital, Hässleholm, Skåne County
  - Department of Orthopedics - Skåne University Hospital Malmö, Malmo, Skåne County
  - Capio Ortho Center, Malmo, Skåne County
  - Capio Ortho Center Göteborg, Gothenburg, Västra Götaland County
  - Department of Orthopedics - Eksjö Hospital, Eksjö
  - Department of Orthopedics - Falun Hospital, Falun
  - Department of Orthopedics - Sahlgrenska University Hospital, Mölndal
  - Department of Orthopedics - Östersund Hospital, Östersund
  - Department of Orthopedics - Uppsala University Hospital, Uppsala
  - Department of Orthopedics - Växjö, Vaxjo

IPD SHARING:
Plan to Share IPD: No
We plan to publish the results of our findings in a scientific journal. Data will be published on a population level and no IPD will be shared with other researchers.

REFERENCES:
- [Background] Ellis SJ, Yu JC, Williams BR, Lee C, Chiu YL, Deland JT. New radiographic parameters assessing forefoot abduction in the adult acquired flatfoot deformity. Foot Ankle Int. 2009 Dec;30(12):1168-76. doi: 10.3113/FAI.2009.1168. PMID 20003875
- [Background] Iossi M, Johnson JE, McCormick JJ, Klein SE. Short-term radiographic analysis of operative correction of adult acquired flatfoot deformity. Foot Ankle Int. 2013 Jun;34(6):781-91. doi: 10.1177/1071100713475432. Epub 2013 Feb 5. PMID 23386748
- [Background] Jordan TH, Rush SM, Hamilton GA, Ford LA. Radiographic outcomes of adult acquired flatfoot corrected by medial column arthrodesis with or without a medializing calcaneal osteotomy. J Foot Ankle Surg. 2011 Mar-Apr;50(2):176-81. doi: 10.1053/j.jfas.2010.12.008. PMID 21354002
- [Background] Mattesi L, Ancelin D, Severyns MP. Is subtalar arthroereisis a good procedure in adult-acquired flatfoot? A systematic review of the literature. Orthop Traumatol Surg Res. 2021 Oct;107(6):103002. doi: 10.1016/j.otsr.2021.103002. Epub 2021 Jun 30. PMID 34216843
- [Background] Mercun A, Kovacic B, Suhodolcan L, Drobnic M. Patient Outcomes Following Extra-Osseous Talo-Tarsal Stabilization for Foot Hyperpronation. J Foot Ankle Surg. 2022 Mar-Apr;61(2):318-322. doi: 10.1053/j.jfas.2021.09.002. Epub 2021 Sep 9. PMID 34600818
- [Background] Myerson MS, Badekas A, Schon LC. Treatment of stage II posterior tibial tendon deficiency with flexor digitorum longus tendon transfer and calcaneal osteotomy. Foot Ankle Int. 2004 Jul;25(7):445-50. doi: 10.1177/107110070402500701. PMID 15319100
- [Background] Osbeck I, Coster M, Montgomery F, Atroshi I. Surgically treated adult acquired flatfoot deformity: Register-based study of patient characteristics, health-related quality of life and type of surgery according to severity. Foot Ankle Surg. 2023 Jun;29(4):367-372. doi: 10.1016/j.fas.2023.03.003. Epub 2023 Mar 15. PMID 36948921
- [Background] Ozan F, Dogar F, Gencer K, Koyuncu S, Vatansever F, Duygulu F, Altay T. Symptomatic flexible flatfoot in adults: subtalar arthroereisis. Ther Clin Risk Manag. 2015 Oct 16;11:1597-602. doi: 10.2147/TCRM.S90649. eCollection 2015. PMID 26527876
- [Background] Reilingh ML, Beimers L, Tuijthof GJ, Stufkens SA, Maas M, van Dijk CN. Measuring hindfoot alignment radiographically: the long axial view is more reliable than the hindfoot alignment view. Skeletal Radiol. 2010 Nov;39(11):1103-8. doi: 10.1007/s00256-009-0857-9. Epub 2010 Jan 9. PMID 20062985
- [Background] Saxena A, Via AG, Maffulli N, Chiu H. Subtalar Arthroereisis Implant Removal in Adults: A Prospective Study of 100 Patients. J Foot Ankle Surg. 2016 May-Jun;55(3):500-3. doi: 10.1053/j.jfas.2015.12.005. Epub 2016 Feb 11. PMID 26874830
- [Background] Viladot Voegeli A, Fontecilla Cornejo N, Serra Sandoval JA, Alvarez Goenaga F, Viladot Perice R. Results of subtalar arthroereisis for posterior tibial tendon dysfunction stage IIA1. Based on 35 patients. Foot Ankle Surg. 2018 Feb;24(1):28-33. doi: 10.1016/j.fas.2016.10.006. Epub 2016 Nov 5. PMID 29413770
- [Background] Walley KC, Greene G, Hallam J, Juliano PJ, Aynardi MC. Short- to Mid-Term Outcomes Following the Use of an Arthroereisis Implant as an Adjunct for Correction of Flexible, Acquired Flatfoot Deformity in Adults. Foot Ankle Spec. 2019 Apr;12(2):122-130. doi: 10.1177/1938640018770242. Epub 2018 Apr 12. PMID 29644885